CLINICAL TRIAL: NCT03575611
Title: Definitive Radiation-Based Treatment Strategy for Oligometastatic and Low Metastatic Burden Renal Cell Carcinoma in Lieu of Systemic Therapy
Brief Title: Stereotactic Body Radiation Therapy in Treating Patients With Oligometastatic Renal Cell Carcinoma
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: PI Request
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018-0203; NCI-2018-01083 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2018-0203 (Other: M D Anderson Cancer Center); P30CA016672 (NIH)
Record Dates: First submitted 2018-06-20; First posted 2018-07-02 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-10

CONDITIONS: Metastatic Renal Cell Carcinoma; Stage IV Renal Cell Cancer AJCC v8
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Biopsy; Specimen Handling; Magnetic Resonance Spectroscopy; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (SBRT) (Experimental): Patients undergo SBRT over 1 day to 3 weeks based on the judgment of the treating radiation oncologist. If the disease spreads to a new lesion that can be treated with local therapy, patients may repeat SBRT over 1 day to 3 weeks based on the judgment of the treating radiation oncologist. Patients may undergo blood sample collection throughout the trial, as well as a tumor biopsy on study. Patients also undergo CT, PET/CT, and/or MRI throughout the trial.
  Interventions: Procedure: Biopsy; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography; Radiation: Stereotactic Body Radiation Therapy

INTERVENTIONS:
Procedure: Biopsy — Undergo tumor biopsy
  Other Names: BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT and/or PET/CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging; PT
Radiation: Stereotactic Body Radiation Therapy — Undergo SBRT
  Other Names: SABR; SBRT; Stereotactic Ablative Body Radiation Therapy

SUMMARY:
This phase II trial studies how well stereotactic body radiation therapy works in treating patients with kidney cancer that has spread to other places in the body (metastatic). Stereotactic body radiation therapy uses special equipment to position a patient and deliver radiation to tumors with high precision. This method may kill tumor cells with fewer doses over a shorter period and cause less damage to normal tissue.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the feasibility definitive radiation therapy (RT) (such as stereotactic body radiation therapy [SBRT]) as a treatment strategy for oligometastatic renal cell carcinoma (RCC) in lieu of systemic therapy.

II. To estimate the progression free survival (PFS) after study enrollment utilizing a strategy of definitive local treatment to all sites of disease in oligometastatic and low metastatic burden RCC as measured by Response Evaluation Criteria in Solid Tumors 1.1 (RECIST 1.1).

III. To determine the systemic therapy free survival after study enrollment

SECONDARY OBJECTIVES:

I. To determine the effect of definitive RT (SBRT) on cellular replication and death, measured by ki-67 staining and others. (Required in Cohort A, but optional in Cohort B) II. To estimate the overall survival at 12 months after study enrollment. III. To estimate the freedom from new lesion development at 12 months. IV. To determine the treatment related toxicities associated with definitive RT as part of definitive local therapy for oligometastatic and low volume metastatic RCC.

EXPLORATORY OBJECTIVE:

I. To determine the association of translational biomarkers including peripheral blood markers and tissue markers with patient outcomes.

OUTLINE:

Patients undergo SBRT over 1 day to 3 weeks based on the judgment of the treating radiation oncologist. If the disease spreads to a new lesion that can be treated with local therapy, patients may repeat SBRT over 1 day to 3 weeks based on the judgment of the treating radiation oncologist. Patients may undergo blood sample collection throughout the trial, as well as a tumor biopsy on study. Patients also undergo computed tomography (CT), positron emission tomography (PET)/CT, and/or magnetic resonance imaging (MRI) throughout the trial.

After completion of study treatment, patients are followed up every 12 weeks for 1 year, and then every 18 weeks thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed diagnosis of RCC of any histology.
* Be willing and able to undergo biopsy of a lesion planned for definitive RT (such as SBRT) both post treatment and pretreatment. If a lesion amenable to definitive RT was biopsied prior to enrollment, this material can be used in lieu of a planned biopsy if the tissue is available for review and ki-67 staining at MD Anderson.

  * Patients may be allowed on this trial without a biopsy if they are deemed medically unfit for biopsy or if the biopsy poses undue risk in the opinion of the treating physician(s).
* Be >= 18 years of age on the day of signing informed consent
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2.

  * NOTE: If subject is unable to walk due to paralysis, but is mobile in a wheelchair, subject is considered to be ambulatory for the purpose of assessing their performance status.
* COHORT A: Oligometastatic RCC patients (=< 5 metastatic lesions at the time of study entry).
* COHORT B: Patients eligible for Cohort A in addition to low volume metastatic patients. Low volume metastatic patients are defined as those with > 5 metastatic lesions, but with =< 5 metastatic lesions when excluding lesions < 1 cm short axis and LNs < 1 cm short axis
* Candidate for definitive local therapy to all sites of active disease per the discretion of the treating physicians
* Absolute neutrophil count (ANC) >= 1,000 /mcL (within 6 weeks prior to study enrollment).
* Platelets >= 50,000 / mcL (within 6 weeks prior to study enrollment).
* Hemoglobin >= 9 g/dL or >= 5.6 mmol/L (within 6 weeks prior to study enrollment).
* Serum total bilirubin =< 1.5 mg//dl (except for subjects with Gilbert syndrome, who may have total bilirubin < 3.0 mg/dl) OR direct bilirubin =< ULN for subjects with total bilirubin levels > 1.5 mg/dl (within 6 weeks prior to study enrollment).
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]) =< 3 X upper limit of normal ULN OR =< 5 X ULN for subjects with liver metastases (within 6 weeks prior to study enrollment).
* At least one site which in the opinion of the treating radiation oncologist is treatable with definitive RT and can be biopsied

Exclusion Criteria:

* Receipt of > 1 line of systemic therapy directed towards the metastatic disease. This exclusion criteria will not apply for Cohort B, including the modified Cohort B definition

  * Systemic therapy as a component of prior definitive therapy directed towards non-metastatic disease will be allowed. For example, patients receiving adjuvant interleukin (IL)-2 after nephrectomy for an initial M0 diagnosis and who subsequently developed metastatic relapse will be allowed on study. In this instance, there will be no mandatory wash-out period required for enrollment.
  * At trial entry the patient must have received their last dose of systemic therapy (e.g. last intravenously [IV] administration of orally [PO] tablet/pill) 4 weeks prior to initiation of the first dose of radiation
* Has a diagnosis of active scleroderma, lupus, or other rheumatologic disease which in the opinion of the treating radiation oncologist precludes safe radiation therapy.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial as determined by the treating physician and/or member of the study team.
* Metastatic effusion (e.g. pleural effusion or ascites). Note that patients with an effusion that is too small to sample will be eligible for the trial.
* Diffuse metastatic processes including leptomeningeal disease, diffuse bone marrow involvement, and peritoneal carcinomatous, which by the discretion of the treating physician cannot be treated definitively.
* Is pregnant or expecting to conceive within the projected duration of the trial at the screening visit.

  * Female subject of childbearing potential should have a negative urine or serum pregnancy within 6 weeks prior to study registration up to the first fraction of radiation.
  * Note: If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2018-06-14 (Actual); Primary Completion 2024-08-20 (Actual); Study Completion 2030-09-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility of incorporating definitive radiation therapy (RT) (such as stereotactic body radiation therapy [SBRT]) into treatment plan for oligometastatic renal cell carcinoma (RCC) in lieu of systemic therapy | Up to 12 months
  Defined as successful completion of all protocol-related treatment with < 7 days of unplanned radiation treatment delays within 3 years of protocol activation.
Feasibility of incorporating definitive RT (such as SBRT) as a treatment strategy for low metastatic burden RCC in lieu of systemic therapy | Up to 12 months
  Defined as successful completion of all protocol-related treatment with < 7 days of unplanned radiation treatment delays within 3 years of protocol approval.
Progression-free survival (PFS) in oligometastatic RCC per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 | At 12 months
  Serial assessment with radiographic imaging will be evaluated. The probabilities of participants remaining alive and progression free will be estimated using the Kaplan Meier method with corresponding 95% confidence intervals.
PFS in low metastatic burden RCC per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 | Up to 12 months
  Serial assessment with radiographic imaging will be evaluated. The probabilities of participants remaining alive and progression free will be estimated using the Kaplan Meier method with corresponding 95% confidence intervals.

SECONDARY OUTCOMES:
Systemic therapy free survival | At 12 months
  The probabilities of patients remaining off systemic therapy at 12 months will be estimated utilizing the Kaplan Meier and model it as a function of potential prognostic factors using Cox proportional hazards regression.
Reduction in cellular replication as measured by ki-67 staining (Cohort A) | Baseline up to 12 months
  The number of cells with ki-67 staining per 10 high powered fields will be calculated in pre- and post SBRT samples. The percent difference in in ki-67 staining will be calculated by dividing the difference in pre- and post- ki67 staining by the pretreatment ki-67. Will estimate the median relative change with 95% confidence interval.
Overall survival | At 12 months
  The probabilities of participants remaining alive will be estimated utilizing the Kaplan Meier method with corresponding 95% confidence intervals.
Freedom from new lesion development | At 12 months
  A participant will be considered to have a new lesion when standard radiographic imaging identifies a new lesion that is non-contiguous with any other lesions measured at baseline. The probabilities of patients remaining free from new lesions will be estimated utilizing the Kaplan Meier method with corresponding 95% confidence intervals.
Treatment related toxicities associated with SBRT | Up to 12 months
  The frequency of grade 2 and higher toxicities attributable to study treatment will be reported for all patients at all follow up visits.

CONTACTS AND LOCATIONS:
Overall Officials: Chad Tang, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Tang C, Sherry AD, Seo A, Hara K, Choi H, Liu S, Sun X, Montoya A, Ludmir EB, Shah AY, Jonasch E, Zurita AJ, Kovitz C, Alhalabi O, Goswami S, Hahn AW, Campbell MT, Hernandez A, Nead KT, Van Loo P, Su S, Battey CJ, LaBella ML, Ratzel S, Acevedo A, Genovese G, Sircar K, Karam JA, Tannir NM, Msaouel P. Metastasis-directed radiotherapy without systemic therapy for oligometastatic clear-cell renal-cell carcinoma: primary efficacy analysis of a single-arm, single-centre, phase 2 trial. Lancet Oncol. 2025 Oct;26(10):1289-1299. doi: 10.1016/S1470-2045(25)00380-8. Epub 2025 Sep 4. PMID 40915303
- [Derived] Tang C, Msaouel P, Hara K, Choi H, Le V, Shah AY, Wang J, Jonasch E, Choi S, Nguyen QN, Das P, Prajapati S, Yu Z, Khan K, Powell S, Murthy R, Sircar K, Tannir NM. Definitive radiotherapy in lieu of systemic therapy for oligometastatic renal cell carcinoma: a single-arm, single-centre, feasibility, phase 2 trial. Lancet Oncol. 2021 Dec;22(12):1732-1739. doi: 10.1016/S1470-2045(21)00528-3. Epub 2021 Oct 28. PMID 34717797